CLINICAL TRIAL: NCT02628548
Title: Neural and Cognitive Changes Associated With Mental Training in Older Adults
Brief Title: Neural Correlates of Successful Cognitive Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2015P001851; R01AG048351 (NIH)
Record Dates: First submitted 2015-11-30; First posted 2015-12-11 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive training program 1 (Experimental): This 8-week program will meet once per week for 1.5 hours. Participants will be trained in performing various cognition enhancing techniques at each class, and will practice these techniques both in class and at home each day for 45 minutes.
  Interventions: Behavioral: Cognitive training program
- Cognitive training program 2 (Experimental): This 8-week program will meet once per week for 1.5 hours. Participants will be trained in performing various cognition enhancing techniques at each class, and will practice these techniques both in class and at home each day for 45 minutes.
  Interventions: Behavioral: Cognitive training program

INTERVENTIONS:
Behavioral: Cognitive training program — 8 week cognitive training program

SUMMARY:
Normal aging is associated with gradual cognitive declines. These mild neurocognitive disturbances affect daily functioning, health status, and quality of life, and likely account for the roughly $2.9 billion lost by the elderly each year to fraud. The goal of this project is to compare two different 8-week training programs to promote successful neural and cognitive aging. Changes in neural structure and cognitive function will be assessed in a cohort of older adults, as well as the long-term stability of these changes over 24 months.

DETAILED DESCRIPTION:
Normal aging is associated with gradual cognitive declines. These mild neurocognitive disturbances affect daily functioning, health status, and quality of life, and likely account for the roughly $2.9 billion lost by the elderly each year to fraud. People are paying millions out of pocket for cognitive training programs like Lumosity to stave off these declines. These cognitive decreases have been strongly associated with normal age-dependent declines in neural structure and function, including cortical thickness decreases (approximately 0.02 mm per decade) across most of the cortical mantle, as well as decreases in the volume of the hippocampus (approximately 1-2% annually), white matter microstructure, and functional connectivity across the brain. Life expectancy is increasing and so identifying interventions that can be widely implemented and that can slow or reverse normal cognitive decline are clinical and public health priorities. Some training programs can improve cognitive performance in cognitively normal older adults, and gains are maintained post training. The investigators hypothesize that different techniques to boost cognition likely works through different neural mechanisms, and thus may provide different cognitive benefits. The goal of this project is to compare two different 8-week training programs to promote successful neural and cognitive aging. Changes in neural structure and cognitive function will be assessed in a cohort of older adults, as well as the long-term stability of these changes over 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 years of age
* Right-handed

Exclusion Criteria:

1. Lifetime history of schizophrenia or psychosis. Any other Axis I diagnosis in the past 12 months.
2. Subjects must not endorse suicidality, homicidality or self-destructive acts or urges as assessed through a structured clinical interview (SCID)
3. History of seizure or significant head trauma (i.e., extended loss of consciousness, neurological sequelae, or known structural brain lesion).
4. Neurological or medical conditions that would interfere with study procedures or confound results, such as conditions that alter cerebral blood flow or metabolism.
5. Use of psychotropic medications within 12 months prior to study.
6. Daily use of any medication that alters neural metabolism or blood flow.
7. Any concurrent psychotherapy.
8. Having taken no more than 8 meditation classes (or related practices such as yoga, Tai Chi, or Chi Gong) of any kind in the past 6 months, or more than 15 classes in the past 12 months.
9. Pregnancy.
10. Metallic implants or devices contraindicating magnetic resonance imaging.
11. Claustrophobia

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in brain structure | 8 weeks
  Gray matter structure will be assessed before and after the 8 week programs.
Change in brain activity during a memory test | 8 weeks
  Brain activity during a memory task will be assessed before and after the 8 week programs.

SECONDARY OUTCOMES:
Blood markers | baseline, 8 weeks, 12 and 24 months
  Blood will be collected at baseline, 8 weeks, 12 and 24 months. This will be used to assess changes in various biomarkers that are known to change with aging.
Change in cognition | 2 years
  Participants will complete a series of memory and attention tests at 6 time-points: baseline, 2 months, 6 months, 12 months 18 months and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sevinc G, Rusche J, Wong B, Datta T, Kaufman R, Gutz SE, Schneider M, Todorova N, Gaser C, Thomalla G, Rentz D, Dickerson BD, Lazar SW. Mindfulness Training Improves Cognition and Strengthens Intrinsic Connectivity Between the Hippocampus and Posteromedial Cortex in Healthy Older Adults. Front Aging Neurosci. 2021 Aug 27;13:702796. doi: 10.3389/fnagi.2021.702796. eCollection 2021. PMID 34512305